CLINICAL TRIAL: NCT04648072
Title: Total Regional Anesthesia Techniques Resulting in up and Early Discharge Following Knee Surgery: An Opioid Reduction Plan for Transitional Pain at Home.
Brief Title: How Does the Addition of Adductor Canal Block to Local Infiltration Affect Recovery in Patients Undergoing Total Knee Arthroplasty? A Feasibility Study.
Acronym: TRUE KnORTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Sciences North Research Institute (Other)
Collaborators: Dedicated Anesthesia Research Enhancement Grant (Unknown)
Responsible Party: Principal Investigator, Kim Wong, Principal Investigator, Northern Ontario School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRUE KnORTH
Record Dates: First submitted 2020-11-09; First posted 2020-12-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis; Arthritis Knee; Knee Disease; Opioid Use
Keywords: Quality of Recovery-15 Survey; Peripheral Nerve Block; Local Infiltration; Adductor Canal Block; Periarticular Injection; Regional Anesthesia; Total Knee Arthroplasty; Orthopedics; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized control trial. Two arms of 30 participants will be included in this study. The experimental arm will receive both the periarticular injection and the adductor canal block with local anesthetic, while the control group will receive the periarticular injection and a sham adductor canal block with normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periarticular Injection + Adductor Canal Block (Local Anesthestic) (Experimental): The experimental arm with receive both the periarticular injection and the adductor canal block.
  The periarticular injection will be performed by the surgeon and will consist of 100 mL of injectate being distributed in the following manner: 30 mL to the posterior capsule, 10 mL to the medial collateral ligament, 10mL to the lateral collateral ligament (ensuring not to infiltrate common peroneal nerve), 20mL to the quadriceps and anterior capsule, and 30 mL to the subcutaneous tissue. The periarticular injection will consist of 250 mg of ropivacaine, 30 mg of ketorolac, and 0.5 mg of epinephrine.
  The adductor canal block will be completed by the anesthesiologist after spinal anesthesia has been initiated, but before the surgery commences. The block will be completed using an aseptic technique under dynamic, in-plane US guidance. 20 mL of injectate consisting of 100mg of ropivicaine and 50 mcg of epinephrine will be injected around the hyperechoic saphenous nerve.
  Interventions: Procedure: Adductor Canal Block; Procedure: Periarticular Injection
- Periarticular Injection + Adductor Canal Block (Normal Saline) (Placebo Comparator): The control arm with receive a periarticular injection and a sham adductor canal block.
  The periarticular injection will be carried out in the same manner as described for the experimental group. The technical aspects of the sham adductor canal block will be the same as for the experimental arm; however, the injectate will consist of 20 mL of normal saline.
  Interventions: Procedure: Adductor Canal Block; Procedure: Periarticular Injection

INTERVENTIONS:
Procedure: Adductor Canal Block — As previously described.
Procedure: Periarticular Injection — As previously described.

SUMMARY:
The use of periarticular injection and adductor canal block are well-established techniques used both in combination or in isolation in the management of postoperative pain for patients undergoing total knee arthroplasty. The aim of this study is to investigate whether combining these two techniques have an added benefit, compared to periarticular injection alone, with respect to quality of recovery, functional return, discharge readiness, and short and long term post-operative narcotic use.

DETAILED DESCRIPTION:
This study is a double blinded, randomized control trial. In order to create a blinded study, each participant will receive two injections; a single shot adductor canal block (ACB) and a periarticular injection (PI). All syringes will be non-identifiable to the surgeon, anesthetist and the patient.

Specifically, the two arms are:

Arm 1: PI (Ropivacaine + Ketorolac + Epinepherine) + ACB (Ropivacaine)

Arm 2: PI (Ropivacaine + Ketorolac + Epinepherine) + ACB (Normal Saline)

The aim of this study is to investigate whether combining these two techniques have an added benefit, compared to periarticular injection alone. The investigators hypothesize that the addition of an adductor canal block will translate to a superior quality of recovery, as well as an improvement in functional return, discharge readiness and less short-term and long-term post-operative narcotic use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring primary total knee arthroplasty
2. Patients interested in being part of the study
3. Eligible to receive spinal anesthesia

Exclusion Criteria:

1. Age < 18 years
2. BMI > 40 kg/m2
3. Deemed unsuitable for regional anesthesia
4. Planned general anesthesia
5. Hepatic insufficiency/Intolerance to acetaminophen
6. Renal insufficiency (defined by eGFR <60)
7. Chronic opioid use (individuals requiring the equivalent of 1 mg or more of intravenous morphine, or 3 mg or more of oral morphine, per hour for greater than 1 month)
8. Sulpha allergy
9. Allergy or intolerance to trial medications
10. Clinical Frailty Scale Score > 4
11. Surgery scheduled on a weekend

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Scoring on the Quality of Recovery-15 Survey | Up to 4 weeks post-operatively.
  The Quality of Recovery-15 Survey is a validated patient-reported outcome questionnaire that measures the quality of recovery after surgery and anaesthesia. The 11-point numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery). To be completed pre-operatively, and on POD#1, POD#10, and POD#28.
Feasibility Outcomes | End of project
  Defined by eligibility, recruitment rate, adherence to intervention protocol, percentage of completed outcome measures, participant retention

SECONDARY OUTCOMES:
Postoperative Pain | Throughout hospital stay, an average of 1-2 days.
  Pain will be assessed using the numeric rating scale (NRS) - an eleven point scale from 0 (no pain) to 10 (worst pain imaginable) - at rest and with movement. To be completed twice daily while in hospital.
Range of Motion | Throughout hospital stay, an average of 1-2 days.
  To be assessed by physiotherapy personnel twice daily while in hospital.
Time to Meet Discharge Criteria | Throughout hospital stay, an average of 1-2 days.
  Discharge criteria will be assessed by physiotherapy personnel and will include the ability to transfer in and out of bed independently, the ability to transfer on and off the toilet independently, the ability to ambulate independently with or without an assistive device for 50 meters, and the ability to do stairs if they are present in the patient's home environment. Time to meet discharge will be reported in half days. To be completed twice daily while in hospital.
Narcotic Consumption | Up to 4 weeks post-operatively.
  In hospital opioid consumption will be recorded and tracked by nursing personnel and will be assessed twice daily while in hospital. Post-discharge opioid consumption will be assessed using a questionnaire that will be administered by the Research Assistant over the phone. Corroboration of patient report will be completed by the Pharmacy Department. Post-discharge opioid consumption will be tracked on POD #10 and POD#28.
Timed Up and Go (TUG) Test | Throughout hospital stay, an average of 1-2 days.
  To be assessed by physiotherapy personnel twice daily while in hospital.

OTHER OUTCOMES:
Opioid-Related Side Effects (Vomiting & Pruritus) | Throughout hospital stay, an average of 1-2 days.
  Both vomiting and pruritic events will be assessed by nursing personnel daily while in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wong, M.D., Principal Investigator — Health Sciences North
Locations (1):
- Health Sciences North, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No